CLINICAL TRIAL: NCT04488965
Title: Study of the Therapeutic Effects of Cortical Autograft Implantation in Patients With Cerebral Ischemia
Acronym: AVCell
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Associate professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVCell2020
Record Dates: First submitted 2020-06-02; First posted 2020-07-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Ischemic Stroke
Keywords: autologous transplant; brain cell therapy; motor cortex lesion; cortical autograft
MeSH Terms: conditions — Ischemic Stroke | interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: monocentric, non-randomized, open-label with single-arm design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous neural cell ecosystems - ANCE (Experimental): The patient will undergo first surgery under general anesthesia for the collection of the cortical biopsy (5x5x5 mm biopsy of non-dominant frontal cortex). After the production of ANCE from the cortical biopsy, which last 8 to 12 weeks, the patient will undergo a second neurosurgery, for the stereotaxic reimplantation of ANCE under general anesthesia.
  Interventions: Other: Autologous transplant

INTERVENTIONS:
Other: Autologous transplant — Autologous transplant obtained from cortical biopsy

SUMMARY:
Brain lesions in the adult have dramatic consequences, because the spontaneous capacity of the brain to functionally recover is limited. Besides existing rehabilitative therapeutic approaches (e.g. physiotherapy), several lines of research aim at developing treatments to promote and refine brain plasticity to enhance functional recovery following brain injury.

This pilot clinical study aims at enrolling subjects victim of a stroke with neuronal destruction leading to a disabling motor deficit. Usually these patients benefit from intensive neurorehabilitation which allows them to progress up to a certain point but when their recovery plateau is reached; current medicine is disarmed and no effective treatment allows, to date, to improve further their performance. This monocentric pilot study aims at evaluating the feasibility and safety of Autologous Neural Cell Ecosystems (ANCE), which is a cortical autograft intended to be used on stroke patients, for the replacement of motor neurons destroyed during an ischemic stroke.

DETAILED DESCRIPTION:
Using neural grafts to restore function after lesions of the central nervous system is a challenging strategy. Most of the transplantation experience acquired the last decades was focused on fetal neuronal grafts. However, despite the great enthusiasm generated by this approach, ethical controversies, immune rejection, and lack of fetal donors remain a major problem. Therefore, autotransplantation of adult brain cells represents an attractive restoration alternative to bypass the caveats of fetal grafting.

The optimization of the procedure to obtain ANCE, a cortical autograft obtained from cortical biopsy, was first successfully demonstrated in producing long-term primary culture of adult human brain cells from temporal lobe tissues obtained from epilepsy and trauma neurosurgical patients. ANCE has been characterized as an ecosystem of autologous neural cells in suspension, composed of several cell types: astrocytes, proliferative progenitors and quiescent progenitors.

The production of ANCE has been implemented to prepare long-term primary culture from primate cortical biopsies. This allowed assessing the feasibility of autotransplantation from brain biopsy to reimplantation of cultured brain cells in a non-human primate model of motor cortex lesion. On the same model of cerebral cortex lesion in nonhuman primates, further study demonstrated, by quantitative behavioral evidence, the beneficial outcome of cell therapy following injury of the cerebral cortex.

Based on the encouraging results from past experiences on non-human primate model of motor cortex lesion, this monocentric pilot study aims at evaluating the feasibility and safety of ANCE (Autologous Neural Cell Ecosystems), which is cortical autograft intended to be used on stroke patients, for the replacement of motor neurons destroyed during an ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 75 years old.
* Victim of a first ischemic stroke in superficial Sylvian territory with at least frontal damage.
* Cerebral ischemic lesion demonstrated by MRI.
* Stroke older than one year.
* Presence of a motor hemi-syndrome with at least one involvement of the upper limb.
* Stable neurological deficit in motor function of the limb greater than two months apart before enrolling the patient in the study.
* Woman of childbearing potential with a negative blood pregnancy test before the biopsy and using a reliable method of contraception during the study.
* Patient capable of discernment and of giving informed consent himself.
* Absence of other serious pathologies or comorbidities.

Exclusion Criteria:

* Brain lesions or a history of stroke or brain hemorrhage.
* Signs of peripheral neurological damage, such as radicular or trunk involvement
* History of spinal cord problems.
* History of neurosurgical intervention in the brain.
* surgical intervention contraindications.
* Anticoagulation, if it cannot be interrupted one week before and one week after each of the 2 brain surgeries.
* Coagulation disorders.
* Treatment of botulinum toxin during the last 3 months before inclusion.
* Seizures or anti-epileptic treatment.
* Global cognitive disorders, such as degenerative or vascular dementia.
* High blood pressure difficult to control.
* Alcohol or drug abuse.
* Known neoplasia.
* Inability to understand or cooperate in the study.
* MRI contraindication
* Pregnancy
* Penicillin intolerance or allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility and safety of ANCE treatment by evaluating the incidence of treatment-related adverse events | 54 months (Visits will be carried out 2 years and 4 years after reimplantation in order to ensure that there is no long-term complication of ANCE reimplantation)
  Successful collection of the cortical biopsy; in vitro production of the cortical autograft from the cortical biopsy; and reimplantation of the transplant without treatment-related serious adverse events.

SECONDARY OUTCOMES:
Change in the medium term of the participant score when assessing the "Catherine Bergego Scale" (CBS) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  CBS is an observational, functional, performance based assessment, being 0 (indicating no neglect) to 30 (indicating severe neglect).
Change in the medium term of the participant score when assessing the NIHSS | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  NIHSS quantifies the impairment caused by a stroke, being 0 no stroke symptoms, and 42 severe impairment.
Change in the medium term of the participant score when assessing the Modified Rankin Scale | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  The Modified Rankin Scale measures the degree of disability or dependence in the daily activities, being 0 no symptoms, 5 severe disability and 6 dead.
Change in the medium term of the patient score when assessing the Action Research Arm Test (ARAT) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  ARAT assesses upper limb functioning using observational methods (19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement)), being 0 incapability to perform the test, and 57 being able to perform the test normally.
Change in the medium term of the patient score when assessing the Box and Block Test (BBT) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  BBT measures unilateral gross manual dexterity. The BBT is composed of a box divided in two compartments by a partition and 150 blocks. Participants are scored based on the number of blocks transferred from one compartment to the other compartment in 60 seconds. Higher scores are indicative of better manual dexterity.
Change in the medium term of the patient score when assessing the Resistance to passive movement scale (Repas) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  Assessed for the upper limb and lower limb (maximum score being 56 and 48, respectively, being 0 no increase in muscle tone and the maximum score increased resistance to passive movement (affected part rigid in flexion or extension).
Change in the medium term of the patient score when assessing Activities of Daily Living (ADL) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  Activities of Daily Living (ADLs) are tasks related to personal care: for each task the score varies from 7 when completely independent, to 1 when requiring total support. Hence, higher scores are indicative of better functional independence.
Change in the medium term of the patient score when assessing Rivermead Mobility Index | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  The Rivermead Mobility Index is a measure of disability related to bodily mobility. It demonstrates the patient's ability to move her or his own body, being 0 the lowest score and 15 the highest. The highest the score the better the mobility.
Change in the medium term of the patient score when assessing Berg Balance Scale | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of 14 predetermined tasks. Score ranges from 0 to 4 for each task, being the highest total score 56, i.e. completely independent.
Change in the medium term of the patient score when assessing London Handicap Scale (LHS) | up to 54 months (Assessment is performed at each visit up to the last visit 4 years after reimplantation)
  The London Handicap Scale can be used to determine the effect of chronic disorders on a person's functional ability using a self-completion questionnaire. Minimum scale value is 0 and maximum is 1, with 1 indicating normal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland